CLINICAL TRIAL: NCT07113379
Title: Study for Prevention of Cervical Cancer in Spain
Acronym: REVIVE
Status: Not yet recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: REVIVE
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer Screening; HPV Vaccination
MeSH Terms: interventions — Papillomavirus Vaccines; Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Evaluate the effectiveness of current Human Papillomavirus (HPV) vaccination and screening programs in reducing cervical cancer incidence in Spain. — Data will be collected from existing medical records and supplemented with a specific questionnaire administered to the participating patients.

SUMMARY:
The REVIVE study aims to analyze the current status of Human Papillomavirus (HPV) vaccination programs and cervical cancer screening strategies in Spain. Its objective is to gain a comprehensive understanding of the effectiveness of these preventive measures, as well as to identify the main barriers to access and the existing inequalities in care. The study will also examine the impact of misinformation on population engagement and on the overall equity of the prevention system.

Despite significant advances in both vaccination and screening efforts, cervical cancer remains a major public health concern in Spain. In 2024 alone, 2,259 new cases were diagnosed, that incidence has remained relatively stable in recent years, even decades. Mortality rates have also shown little change, with over 600 deaths annually, totaling nearly 10,000 in the last 15 years.

To address this, the study plans to include approximately 200 patients diagnosed with cervical cancer in Spain between 2019 and 2024. It is a retrospective, observational, and non-interventional study. Data will be collected from existing medical records and supplemented with a specific questionnaire administered to the participating patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix.
* Diagnosis established between 2019 and 2024.

Exclusion Criteria:

* Patients aged below 18 years at diagnosis.
* Diagnosis of other cervical cancer histologies (e.g., neuroendocrine tumors, sarcoma, lymphoma).
* Patents with significant cognitive impairment precluding informed consent for data utilization, where applicable.
* Patients with incomplete medical records relevant to the study variables.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV vaccination and cervical cancer screening among patients diagnosed with cervical cancer in Spain | 2019-2024
  Proportion of individuals diagnosed with cervical cancer who have previously received the HPV vaccine and/or undergone cervical cancer screening prior to their cervical cancer diagnosis. The objective is to assess the effectiveness of national prevention strategies, identify gaps in vaccine and screening coverage, and understand potential barriers to early detection and vaccination.

SECONDARY OUTCOMES:
Percentage of HPV vaccination and screening coverage by region and demographic factors | 2019-2024
  This objective aims to determine the proportion of individuals who have received HPV vaccination and/or undergone cervical cancer screening, stratified by geographic region and key demographic factors such as age and ethnicity. The goal is to identify disparities in preventive healthcare access.
Association between misinformation and socioeconomic factors and the rate of HPV vaccination and screening | 2019-2024
  This objective seeks to evaluate how misinformation and socioeconomic factors (income level, education, employment status, and healthcare access) influence the rates of HPV vaccination and participation in cervical cancer screening programs.
Reported frequency and nature of barriers to accessing to HPV vaccination and cervical cancer screening | 2019-2014
  This objective aims to identify and categorize the most commonly reported barriers that individuals face when trying to access to HPV vaccination and screening programs.